CLINICAL TRIAL: NCT05751928
Title: A Randomized Study of the Efficacy and Safety of Neoadjuvant Therapy With BCD-217 (Nurulimab + Prolgolimab) Versus Standard Adjuvant Therapy With Pembrolizumab in Patients With Resectable Stage III Skin Melanoma.
Brief Title: A Study of Neoadjuvant Therapy With BCD-217 (Nurulimab + Prolgolimab) in Patients With Resectable Stage III Skin Melanoma
Acronym: NEO-MIMAJOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCD-217-3
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Melanoma Stage III; Melanoma (Skin)
Keywords: PD-1; CTLA-4; prolgolimab; nurulimab; immunotherapy; checkpoint inhibitors; CPI; programm death; cytotoxic T-lymphocyte-associated protein; Neoadjuvant Melanoma; Adjuvant Melanoma
MeSH Terms: conditions — Melanoma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects with pCR and pnCR (Group 1A) (Experimental): Subjects will receive 2 cycles of BCD-217 neoadjuvant therapy, followed by index lymph node removal.
  Subjects with pathological complete (pCR) and near complete response (pnCR) (Group 1A): excision of the primary lesion (if not previously performed) without regional lymphadenectomy, followed by up to 12 months of anti-PD1 agent in the adjuvant setting.
  Interventions: Biological: BCD-217; Biological: anti-PD1; Procedure: Excision of the primary lesion
- Subjects with a pPR or pNR to neoadjuvant therapy (Group 1B) (Experimental): Subjects will receive 2 cycles of BCD-217 neoadjuvant therapy, followed by index lymph node removal.
  Subjects with a pathological partial response (pPR) or non-responders (pNR) to neoadjuvant therapy (Group 1B): excision of the primary lesion (if not performed earlier), regional lymphadenectomy, then up to 12 months of adjuvant therapy with anti-PD1 agent.
  Interventions: Biological: BCD-217; Biological: anti-PD1; Procedure: Excision of the primary lesion; Procedure: Regional lymphadenectomy
- Control Group (Group 2) (Active Comparator): Subjects start treatment with excision of the primary lesion (if not previously performed), regional lymphadenectomy followed by adjuvant therapy with anti-PD1 agent (up to 12 months). This approach is considered the standard therapy for patients in the target population.
  Interventions: Procedure: Excision of the primary lesion; Procedure: Regional lymphadenectomy

INTERVENTIONS:
Biological: BCD-217 — BCD-217 (anti-CTLA4 agent nurulimab + anti-PD1) once every 3 weeks in the neoadjuvant setting
  Other Names: nurulimab+prolgolimab
  Arms: Subjects with a pPR or pNR to neoadjuvant therapy (Group 1B); Subjects with pCR and pnCR (Group 1A)
Biological: anti-PD1 — anti-PD1 agent in the adjuvant setting
  Arms: Subjects with a pPR or pNR to neoadjuvant therapy (Group 1B); Subjects with pCR and pnCR (Group 1A)
Procedure: Excision of the primary lesion — Excision of the primary lesion will be performed per standard of care.
Procedure: Regional lymphadenectomy — Regional lymphadenectomy will be performed per standard of care.
  Arms: Control Group (Group 2); Subjects with a pPR or pNR to neoadjuvant therapy (Group 1B)

SUMMARY:
This study is an open-label, randomized, comparative phase III study, which will include subjects with resectable stage III skin melanoma (up to 3 resectable transient metastases are acceptable).

DETAILED DESCRIPTION:
In both study groups, adjuvant therapy is possible until melanoma progresses to unresectable stage III-IV, unacceptable toxicity, withdrawal of ICF or the end of the therapy period (12 months).

In case of postoperative relapse of the disease, at the decision of the investigator and if the lesion is resectable, radical surgical treatment can be carried out (R0 - resection) in accordance with current clinical guidelines without withdrawing the patient from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and the subject's ability to comply with the requirements of the clinical study protocol;
2. Age ≥ 18 years at the time of signing the informed consent form;
3. Histologically or cytologically confirmed (documented results of relevant studies are available) resectable stage IIIB/C/D skin melanoma;
4. At least one clinically detectable lymph node accessible for biopsy and not more than three resectable in-transit metastases .

   Clinically detectable lymph nodes include:
   * Palpable lymph nodes with pathologically confirmed melanoma
   * Non-palpable but enlarged (≥15 mm in smallest diameter, RECIST 1.1) lymph nodes with pathologically confirmed melanoma
5. Subject's consent to a biopsy;
6. Consent to the evaluation of the PD-L1 status and BRAF V600 mutation status ;
7. ECOG score 0-1;
8. Life expectancy of at least 5 years;
9. Willingness of subjects and their sexual partners of childbearing potential to use reliable methods of contraception from the date of signing the informed consent form throughout the study period and for 24 weeks after the administration of the last dose of the investigational therapy.

Exclusion Criteria:

1. Ocular melanoma;
2. Mucosal melanoma;
3. Distant metastases;
4. Impossibility of radical resection of the tumor, metastasis and/or involved lymph nodes;
5. Presence of only in-transit transit/satellite metastases without confirmed involvement of lymph nodes;
6. Prior therapy with checkpoint inhibitors (e.g. anti-CTLA-4 and/or anti-PD-1/PD-L1/PD-L2 products);
7. Prior therapy with BRAF and MEK protein kinase inhibitors;
8. Prior radiation therapy;
9. Inability to determine BRAF status;
10. Subjects with severe comorbidities, with life-threatening acute complications of the underlying disease at the time of signing the informed consent form;
11. Current concomitant diseases at the time of screening, which increase the risk of severe adverse events during surgery and/or study therapy administration;

    * stable angina, functional class III-IV;
    * unstable angina or a history of myocardial infarction within less than 6 months prior to signing the informed consent form;
    * moderate to severe cardiac failure (NYHA classes III and IV);
    * uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg) ;
    * a history of atopic asthma , angioneurotic edema;
    * respiratory failure (moderate to severe), grade 3 or 4 chronic obstructive pulmonary disease;
    * any other concomitant diseases (including, but not limited to, metabolic, hematological, renal, hepatic, pulmonary, neurological, endocrine, cardiac, infectious, gastrointestinal disorders), which expose the subject to an unacceptable risk during surgery or study therapy;
12. Known or suspected systemic autoimmune diseases (including, but not limited to, systemic lupus erythematosus, Crohn's disease, ulcerative colitis (UC), systemic scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome, etc.) ;
13. A history of interstitial pulmonary disease or pneumonitis requiring systemic glucocorticoids;
14. The need for glucocorticoid therapy (at >10mg/day prednisolone equivalent doses) or any other drugs with immunosuppressive effects within 6 months prior to randomization;
15. Use of immunostimulants, monoclonal antibodies and/or colony-stimulating factors within less than 4 weeks prior to randomization in the study;
16. Hematological abnormalities :

    * neutrophils <1.5×109/L;
    * platelets <100×109/L;
    * hemoglobin <90 g/L;
17. Renal impairment: creatinine ≥1.5×ULN;
18. Hepatic impairment :

    * Total bilirubin ≥1.3×ULN (except for subjects with Gilbert's syndrome, in whom bilirubin levels should not exceed 50 μmol/L);
    * ALP, AST or ALT ≥1.5×ULN;
19. Any surgery within less than 28 days prior to randomization in the study;
20. History of oncological disease, except for radically treated diseases with remission for over 5 years prior randomization in this study ;
21. Conditions limiting the subject's ability to comply with the Protocol requirements (in the Investigator's opinion );
22. Participation in other clinical studies within less than 30 days prior to randomization and during this clinical study ;
23. Acute infections or activation of chronic infectious diseases or systemic antibacterial therapy within less than 28 days prior to randomization;
24. Active hepatitis B, active hepatitis C (confirmed by PCR), HIV-infection, currently or previously ;
25. Impossibility to administer the investigational product intravenously;
26. Impossibility to administer intravenous contrast agents (including due to hypersensitivity to contrast media);
27. Hypersensitivity to any of the components of BCD-217, prolgolimab or pembrolizumab;
28. A history of hypersensitivity to monoclonal antibody products;
29. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
event free survival (EFS) | 24 months

SECONDARY OUTCOMES:
overall survival (OS) | 24 months
distant metastases-free survival (DMFS) | 24 months
pathologic response rate (pRR) | 24 months
The proportion of subjects with treatment-related adverse events; | 24 months
The proportion of subjects experiencing any grade 3 or higher adverse events | 24 months
The proportion of subjects with SAEs | 24 months
The proportion of subjects with immune-related adverse events of any severity | 24 months
The proportion of subjects with severe immune-related adverse events (grade 3 or higher according to CTCAE v.5.0) | 24 months
The proportion of subjects requiring treatment discontinuation due to AEs | 24 months
The proportion of BAb and NAb positive subjects | 24 months

CONTACTS AND LOCATIONS:
Locations (36):
- Belarus (4):
  - State Institution "Republican Scientific and Practical Center of Oncology and Medical Radiology named after A.I. N.N. Alexandrov", Lesnoy
  - Healthcare Institution "Minsk City Clinical Cancer Center", Minsk
  - State Institution "Mogilev Regional Oncological Dispensary", Mogilev
  - Healthcare Institution "Vitebsk Regional Clinical Oncology Center", Vitebsk
- Russia (32):
  - Clinical Oncologic Dispensary No. 1, Krasnodar, Krasnodar Kari
  - Clinical Oncologic Dispensary No. 2, Sochi, Krasnodar Territory
  - Regional Clinical Oncology Hospital, Yaroslavl, Yaroslavl Oblast
  - State Budgetary Healthcare Institution "Chelyabinsk Regional Clinical Center for Oncology and Nuclear Medicine",, Chelyabinsk
  - State budgetary healthcare institution Leningrad Regional Clinical Hospital, Gatchina
  - State Autonomous Health Institution "Republican Clinical Oncology Dispensary of the Ministry of Health of the Republic of Tatarstan named after Professor M.Z. Sigal", Kazan'
  - State budgetary health care institution "Kuzbass clinical oncological dispensary named after M.S. Rappoport", Kemerovo
  - Regional Goverment Budgetary Healthcare State "Kostroma Oncology Center", Kostroma
  - State Budgetary Institution of Healthcare "Leningrad Regional Clinical Oncological Dispensary named after V.I. L.D. Romana", Kuz'molovskiy
  - "Russian Cancer Research Center named after N.N. Blokhin "of the Ministry of Health of the Russian Federation, Moscow
  - Branch of Hadassah Medical LTD Limited Liability Company, Moscow
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - Joint Stock Company "K31 City", Moscow
  - JSC "Medsi Group", Moscow
  - Moscow City Oncology Hospital No. 62, Moscow
  - State budgetary health care institution of the city of Moscow "City Clinical Oncology Hospital No. 1 of the Department of Health of the City of Moscow", Moscow
  - Nizhny Novgorod Region State Budgetary Healthcare Facility "Clinical Diagnostics Center", Nizhny Novgorod
  - LLC "DobroMed", Novosibirsk
  - State Budgetary Healthcare Institution "Novosibirsk Regional Clinical Oncology Center" of the Novosibirsk Region, Novosibirsk
  - Federal State Budgetary Institution "National Medical Research Center for Radiology" of the Ministry of Health of the Russian Federation, Obninsk
  - Budgetary healthcare institution of the Omsk region "Clinical oncological dispensary", Omsk
  - JSC "Modern Medical Technologies", Saint Petersburg
  - Saint-Petersburg Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncological), Saint Petersburg
  - City Hospital #40, Kurortny district, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Saint Petersburg State University", Saint Petersburg
  - Limited Liability Company "American Medical Clinic", Saint Petersburg
  - Limited Liability Company "Oncological Research Center", Saint Petersburg
  - Limited Liability Company "Strategic Medical Systems", Saint Petersburg
  - N.N. Petrov National Medicine Research Center of oncology, Saint Petersburg
  - Private Medical Institution Evromedservis, Saint Petersburg
  - Federal State Educational Institution of Higher Professional Education "Mordovia State University N.P. Ogareva ", Saransk
  - State Health Care Institution "Volgograd Regional Clinical Oncology Dispensary № 1", Volgograd